CLINICAL TRIAL: NCT06394284
Title: IISPT2: Examining 3,4-methylenedioxymethamphetamine (MDMA) Effects on Psychological, Relational and Hyperarousal-Related Neural Reactivity Mechanisms in Veterans With PTSD and MI
Brief Title: Examining 3,4-methylenedioxymethamphetamine (MDMA) Effects on Psychological, Relational and Hyperarousal-Related Neural Reactivity Mechanisms in Veterans With PTSD and Moral Injury
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Herzog Hospital (Other)
Collaborators: Metiv Israel Psychotrauma Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOH_2023-07-02_012787
Record Dates: First submitted 2024-04-07; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: PTSD, Post Traumatic Stress Disorder; Moral Injury
Keywords: MDMA; PTSD; Moral Injury; Oxytocin; veterans; Hyperarousal
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MDMA Assisted Therapy (Experimental): This intensive therapy is comprised of 16 sessions of therapy with two therapists including three long sessions of MDMA assisted therapy followed by an overnight stay and then 3 weekly integration sessions.
  Interventions: Drug: MDMA-AT
- SEA-IT (Experimental): This intensive trauma focused therapy is comprised of 16 sessions of therapy with two therapists including three long sessions of between 6 to 8 hours followed by an overnight stay and then 3 weekly integration sessions. The therapy is modeled on components of Somatic Experiencing, Acceptance and Commitment Therapy and the psychedelic assisted therapy protocols.
  Interventions: Behavioral: SEA-IT

INTERVENTIONS:
Drug: MDMA-AT — As described above in arm description
  Arms: MDMA Assisted Therapy
Behavioral: SEA-IT — As described in arm description
  Arms: SEA-IT

SUMMARY:
Despite being exposed to a high level of potentially traumatic experiences due to exposure to combat, military veterans have poor response rates to traditional PTSD treatments, in some reports, just 1/3 of veterans recover using traditional treatments. In recent years 3,4-methylenedioxymethamphetamine (MDMA), a psychedelic drug has demonstrated a significant treatment potential for severe and treatment resistant PTSD though not specifically in a veteran population. Additionally, even in groups where participants receive a placebo, the effect of the psychedelic treatment formulation, intensive, focused and respectful structure, appears to have promising effects. Indeed, in the current psychedelic literature, the setting and mind with which participant approach psychedelic therapy, significantly contributes to the treatment effect.

The current study proposes to address the major gaps in the theoretical literature by examining the proposed mechanisms by which MDMA enhances the "window of tolerance" for PTSD therapy, specifically in those with comorbid symptoms of moral injury; namely by reducing hyperarousal and enhancing connection (to self and others) and whether MDMA assisted therapy is more successful in reducing PTSD in veterans compared to a matched somatic experiential PTSD treatment, Somatic Experiental Acceptance Intensive Trauma-based therapy, (SEA-IT) which builds upon the promising placebo results, enhancing them with somatic and acceptance based treatment protocols.

DETAILED DESCRIPTION:
Despite being exposed to a high level of potentially traumatic experiences due to exposure to combat, military veterans have poor response rates to traditional PTSD treatments. In recent years 3,4-methylenedioxymethamphetamine (MDMA) has demonstrated a significant treatment potential for severe and treatment resistant PTSD though not specifically in a veteran population. The current study proposes to address the major gaps in the theoretical literature by examining the proposed mechanisms by which MDMA Assisted Therapy (MDMA-AT) enhances the "window of tolerance" for PTSD therapy, specifically in those with comorbid symptoms of moral injury; namely by reducing hyperarousal and enhancing connection (to self and others) and whether MDMA-AT is more successful in reducing PTSD in veterans compared to a matched somatic experiential PTSD treatment (SEA-IT). Sixty male veterans suffering from military-related PTSD, who have participated in at least one attempt at treatment previously, will be randomly assigned (non-blinded) to receive MDMA-AT or somatic-based therapy. All participants will undergo 3 preparation sessions and then three long (8hour) sessions each followed by 3 integration sessions. Hyperarousal will be studied using EEG (electroencephalogram) to detect significant changes in event-related neural responses and cortisol responsivity to treatment. Additionally measures of PTSD symptoms of hyperarousal and a specific measure of emotion regulation abilities will be studied. Connection will be studied as both mediated by oxytocin responsivity to treatment and as subjective outcome measures of treatment response namely using psychological measures of connection to others and self via interoceptive sensitivity. It is predicted that by using longitudinal modeling and specifically the analysis of mediators of treatment response, the current study will enable both the understanding of the promising effects of MDMA treatment and the refinement of the key contribution of MDMA-AT compared to an intensive, similarly somatic, and experimentally based, non-MDMA treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Were assigned male sex at birth and currently identify as a male (e.g. are not transgender nor taking hormone replacement therapy) 2. Are veterans of the Israeli military 3. Are at least 18 years old. 4. Are fluent in speaking and reading Hebrew 5. Are able to swallow pills. 6. Agree to have EEG (three times) and salivary monitoring (during experimental sessions) at multiple occasions throughout the study.

  7. Agree to have study visits recorded, including Experimental Sessions, Independent Rater assessments, and non-drug therapy sessions.

  8. Must provide a contact (relative, spouse, close friend or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming unwell or unreachable.

  8. Must agree to inform the investigators within 48 hours of any medical conditions and procedures.

  9. Agree to the following lifestyle modifications: comply with requirements for fasting and refraining from certain medications prior to experimental sessions, not enroll in any other interventional clinical trials during the duration of the study, remain overnight at the study site after each experimental Session and be driven home after, and commit to medication dosing, therapy, and study procedures.

Medical History

10. At Screening, meet diagnostic criteria (Diagnostic Statisticians Manual, 5th version, DSM-5) for current military-based PTSD with a symptom duration of 6 months or longer with a history of at least one attempt at psychiatric or psychological treatment.

11. At Screening, have a PCL-5 total score of 33 or greater and at Screening/Baseline a confirmed diagnosis of PTSD per CAPS-5 and a total severity score of 28 or greater.

12. Have a body weight of at least 45 kilograms. Participants with a body weight of 45 to 48 kg must also have a body mass index (BMI) within the range of 18 to 30 kg/m2.

13. Capable of giving signed informed consent.

Exclusion Criteria:

- Medical Conditions

1. Alanine transaminase (ALT) [or aspartate transaminase (AST)]higher than 2 x upper limit of normal (ULN).
2. Total bilirubin higher than 1.5 x ULN (isolated bilirubin higher than; 1.5 x ULN is acceptable if total bilirubin is fractionated and direct bilirubin less than; 35%).
3. Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.

   • Note: Stable chronic liver disease (including Gilbert's syndrome, asymptomatic gallstones, and chronic stable hepatitis B (e.g., the presence of hepatitis B surface antigen or positive hepatitis C antibody test result without evidence of active infection at screening or within 3 months prior to starting study intervention) is acceptable if the participant otherwise meets entry criteria.
4. Have a recent history of clinically significant hyponatremia or hyperthermia.
5. Have a marked baseline QTcF (QT interval corrected for heart rate ) interval higher than 450 ms demonstrated on repeated ECG (electrocardiogram) assessments. Participants whose QTcF exceeds this value during screening may be initially enrolled if a pre-study concomitant medication is suspected to be prolonging the QT-interval. ECGs should be repeated after initial enrollment and tapering off the pre-study concomitant medication to ensure the participant meets eligibility criteria prior to enrolment confirmation and to IMP dosing.

   • Note: The QTcF is the QT interval corrected for heart rate according to Fridericia's formula. It is either machine-read or manually over-read.
6. Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate. This includes, but is not limited to, a history of myocardial infarction, cerebrovascular accident, heart failure, severe coronary artery disease, or aneurysm.

   * Participants with other mild, stable chronic medical problems may be enrolled if the study clinician and Sponsor Investigator (S-I) agree the condition would not significantly increase the risk of MDMA administration or be likely to produce significant symptoms during the study that could interfere with study participation or be confused with side effects of MDMA.
   * Examples of stable medical conditions that could be allowed include but are not limited to human immunodeficiency virus (HIV) infection, gastroesophageal reflux disease (GERD), hypothyroidism (if taking adequate and stable thyroid replacement medication), glaucoma (if approval for study participation is received from an ophthalmologist). Any medical disorder judged by the investigator to significantly increase the risk of harm from MDMA exposure by any mechanism would require exclusion.
7. Have a diagnosis of uncontrolled hypertension, defined as repeated blood pressure readings of ≥140 mmHg systolic or ≥90 mmHg diastolic. The diagnosis may be confirmed by repeated clinic measurements or home blood pressure monitoring if clinically indicated.

   • Participants with well-controlled hypertension that has been successfully treated with anti-hypertensive medicines may be enrolled if they pass a risk assessment and potentially additional screening to rule out underlying cardiovascular disease.
8. Have a history of ventricular arrhythmia at any time, other than occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease.
9. Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
10. Have a history of arrhythmia, other than premature atrial contractions (PACs) or occasional PVCs in the absence of ischemic heart disease, within 12 months of screening.

    • Participants with a history of atrial fibrillation, atrial tachycardia, atrial flutter or paroxysmal supraventricular tachycardia or any other arrhythmia associated with a bypass tract may be enrolled only if they have been successfully treated with ablation and have not had recurrent arrhythmia for at least one year off all antiarrhythmic drugs, as confirmed by a cardiologist.
11. Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).

    Psychiatric Conditions (for MDMA-AT and somatic-based arms)
12. Have engaged in a new form of psychiatric or mental health care within 12 weeks of enrollment, including Electroconvulsive Therapy (ECT), and ketamine-assisted therapy.
13. Are likely, in the investigator's opinion and via observation during the Preparatory Period, to be re-exposed to their index trauma or other significant trauma during the study.
14. Have a current moderate (not in early remission in the 3 months prior to enrollment and meets at least 5 of 11 diagnostic criteria per DSM-5) or severe alcohol or cannabis use disorder within the 12 months prior to enrollment (meets at least 6 of 11 diagnostic criteria per DSM-5).

    • May have current mild alcohol or cannabis use disorder (meets 3 of 11 diagnostic criteria per DSM-5) or moderate alcohol or cannabis use disorder in early remission for the 3 months prior to enrollment (meets 4 or 5 of 11 diagnostic criteria per DSM-5).
15. Have an active illicit drug (other than cannabis) or prescription drug substance use disorder at any severity within 12 months prior to enrollment.
16. Any participant presenting current serious suicide risk, as determined through psychiatric interview, responses to Columbia Suicide Severity Rating Scale (C-SSRS), and clinical judgment of the investigator will be excluded; however, history of suicide attempts is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior, in the judgment of the investigator, will not be enrolled. Any participant presenting with the following on the Baseline/Screening C-SSRS will be excluded:

    * Suicidal ideation score of 4 or greater within the last month of the assessment at a frequency of once a week or more.
    * Suicidal ideation score of 5 within the last 6 months of the assessment.
    * Any suicidal behavior, including suicide attempts or preparatory acts, within the last 6 months of the assessment. Participants with non-suicidal self-injurious behavior may be included if approved by the study clinician.

    Prior/Concomitant Therapy
17. Unable or unwilling to safely taper-off prohibited psychiatric medication with exceptions described in section on Concomitant Medications in study protocol or require use of prohibited medications during experimental sessions.
18. Require use of concomitant medications that could prolong the QT interval during Experimental Sessions.
19. Have used Ecstasy (unregulated material represented as containing MDMA) more than 10 times within the last 10 years, or at least once within 6 months of the first Experimental Session.

    Prior/Concurrent Clinical Study Experience
20. Current enrollment in any other clinical study involving an investigational study treatment or any other type of medical research, unless approved by the study clinician.

    Diagnostic Assessments
21. Have current Personality Disorders assessed via psychiatric assessment (by consultant psychiatrist).
22. Have a current eating disorder with compensatory behaviors
23. Have current major depressive disorder with psychotic features
24. Have a history of, or a current primary psychotic disorder, bipolar affective disorder type 1 or dissociative identity disorder.

    Other Exclusions
25. Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the sponsor-investigator or study clinician, contraindicates participation in the study.
26. Are currently engaged in compensation litigation whereby financial gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders.
27. Lack social support or lack a stable living situation.
28. Previous participation in a MAPS-sponsored MDMA clinical trial.
29. Employees (and their immediate family members) of MAPS, MAPS Public Benefit Corporation, or MAPS Europe B.V; or individuals in a personal relationship with the site investigator.
30. Have any current problem which, in the opinion of the sponsor-investigator or study clinician, might interfere with study participation.

Security Criteria

The current study dealing with intensive treatment of military veterans suffering from PTSD, requires an environment of physical and emotional security for the patients. Safety is critical in the success of the treatment. Since October 7, 2023, we have been in a continuous state of war, which we do not know when it will end. Therefore, we are required at this time to define what security is as a criterion for conducting research at this time, and in relation to the normative reality in the world and in the State of Israel in particular. Therefore:

1. The research will be carried out in Jerusalem and long sessions will not take place when there is a high risk of rocket attack or sirens during the previous day/night.
2. The participants in the study will be military veterans who do not participate or have taken an operational part in the war in the three months prior to the start of their participation in the study.
3. The participants in the study do not have first degree relatives or a partner who are actively serving in a war zone at the time of their participation in the study.
4. The participants live in a permanent and safe place and are not expected to change their place of residence during their participation in the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Identify as male and not taking hormone therapy to transition to female identity
Enrollment: 60 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD | Enrollment and visit 16, two weeks to one month after the final therapy session, approximately 4 months after first visit.
  Clinician-Administered PTSD Scale-5 (CAPS-5) will be performed during the intake interview. The CAPS-5 is a structured clinical interview used to assess the presence of a PTSD diagnosis and PTSD symptom levels over the past month.
Oxytocin | At 4 time points during the 3 long sessions (visit 4, one month after enrollment, visit 8, two months after enrollment and visit 12, three months after enrollment)
  As this study is designated as a mechanisms of change study, the primary outcome is that of exploring the role of oxytocin in the therapeutic process. The primary outcome measure is thus the hormone assessment of increased oxytocin (primary) as mediating the change in PTSD (and MI-exploratory) symptoms. Saliva collection will be the same for both MDMA-assisted and Somatic-based therapy groups and the collection relevant for the measurement of both oxytocin (primary) and cortisol (exploratory). Four saliva samples will be collected at four time points during each of the experimental (or intense) sessions: prior to commencing the session, +90 minutes +210, +320 minutes following the administration of MDMA or commencement of the Somatic-based arm. To assess oxytocin concentrations, saliva samples will be thawed and then dried using a SpeedVac concentrator. The evaporated samples are then reconstituted with an assay diluent. Oxytocin concentrations will be measured using an ELISA kit

SECONDARY OUTCOMES:
Hyperarrousal- EEG | EEG- during visits 3 (three weeks after enrollment), 7 (three weeks after the first long session) and visit 16 (two weeks to a month after the final therapy session) (pre, post 1st long session, post study)
  Mismatch negativity task (MMN) is an event-related potential (ERP) task that examines a pre-attentive brain-response to changes in the acoustic environment (frequent standard tone versus infrequent odd tone).. MMN ERP amplitudes of early N1 components (recorded via scalp-EEG) represent early even-related time-locked difference-waveforms that result from subtracting the standard tone ERP's from the odd-sound ERP's and noting the peak difference in MMN amplitude peak-negativity i.e. MMN amplitudes) around 120 ms after tone-onset. A healthier response is when the infrequent odd sound (change in pitch) produces larger N1 amplitudes (under central prefrontal electrodes) at 100-150 ms post stimulus in comparison to the standard tone early N1 amplitudes, which indicates that automatic "sound-change-detection" registered at auditory and prefrontal cortical networks effectively.
Hyperarrousal- cortisol | Cortisol, as outlined in oxytocin collection
  Cortisol concentrations will be assessed using commercially available ELISA kits (Salimetrics, USA), following the manufacturer's instructions. All samples will be assessed in duplicate.
Moral Injury | visit 1 and visit 16 (two weeks to a month after the final therapy session) (pre-post)
  MIOS- Moral Injury Outcome Scale. Based on over a decades work in the field, a new measure has been designed with promising measurement capabilities though validation work in Israel is ongoing. The Moral Injury Outcome Scale (MIOS) measures shame-related and trust-violation-related outcomes and thus far has demonstrated good discriminative validity between those who have experienced potentially morally injurious events and those who haven't. A higher score indicates higher moral injury.
Functional Impairment | Visits 1,7 (three weeks after first long session),11 (three weeks after second long session) and 16 (two weeks to a month after final therapy session)
  The Sheehan Disability Scale (SDS) is a clinician-rated assessment of functional impairment. The items indicate degree of impairment in the domains of work/school, social life, and home life, with response options based on an eleven-point scale (0=not at all to 10=extremely), and five verbal tags (not at all, mildly, moderately, markedly, extremely). Per FDA request, for participants who are not able to work for reasons related to PTSD, the functional impairment item will be scored as a 10. The SDS takes 1 to 2 minutes to complete.
Self Compassion | Visits 1,7 (three weeks after first long session),11 (three weeks after second long session) and 16 (two weeks to a month after final therapy session)
  The Self Compassion Scale (SCS) is a widely used and widely tested measure of self compassion. If consists of 26 questions measuring the six components of self-compassion: Self-Kindness, reduced Self-Judgment, Common Humanity, reduced Isolation, Mindfulness and reduced Overidentification. The SCS has been validated and factors analyzed with over 11,000 participants and is also in use in current MAPS sponsored studies allowing for data collaboration. Higher scores indicate higher self compassion. Total scores are normally used for research and mean scores for interpretation though there are no clinically validated means (mean scores of 1.0-2.49 are considered to be low, between 2.5-3.5 to be moderate, and 3.51-5.0 to be high). The questionnaire takes around 7 minutes to complete.
Interoception | Visits 1,7 (three weeks after first long session),11 (three weeks after second long session) and 16 (two weeks to a month after final therapy session)
  The Multidimensional Assessment of Interoceptive Awareness 2 (MAIA-2) is a 37 item measure of the ability to notice, be present, not worry, regulate attention to- and trust body experiences. Complementary to the DERS-16, the MAIA-2 focuses on body-related regulation and introspection. It has been used widely in research on mindfulness and compassion based therapies and demonstrated strong relationships to symptom relief and takes around 10 minutes to complete.
Emotional Regulation | Visits 1,7 (three weeks after first long session),11 (three weeks after second long session) and 16 (two weeks to a month after final therapy session)
  The Difficulties in Emotion Regulation Scale-16 question version (DERS-16) is a shortened version of the full Difficulties in Emotion Regulation Scale which is a 36-item self-report questionnaire that measures the extent to which individuals have difficulty responding to distressing emotions. Participants rate items on a 5-point Likert scale (1 = almost never to 5 = almost always) with responses (some reversed) giving a total score in addition to six subscale scores; Awareness, Clarity, Nonacceptance, Impulsivity, Goals, and Strategies. Subscales are scored such that higher scores indicate more difficulties. The shortened version retains the subscales and demonstrates good comparative validity and internal consistency. The subscales of awareness and non-acceptance will be used to assess increased connection to self. The questionnaire takes around 5 minutes to complete.
Attachment | Visits 1,7 (three weeks after first long session),11 (three weeks after second long session) and 16 (two weeks to a month after final sessions.
  Experience of Close Relationships (ECR) Scale is composed of two 18-item subscales measuring attachment anxiety and attachment avoidance, using a 7-point Likert Scale. Subscale scores are obtained by summing and computing the mean and demonstrate high reliability and validity. Scores on this measure will be used as predictive of treatment success with lower anxiety and avoidance predicted to be indicative of better treatment potential and also as a mediator variable of enhanced connection to others (reduction in attachment avoidance). The questionnaire takes around 7 minutes to complete and higher scores indicate higher anxiety or avoidance on subscales.
Attachment | During the three long (visit 4, one month after enrollment, visit 8, two months after enrollment and visit 12, three months after enrollment) and three initial integration sessions (the morning after a long session).
  In addition to overall attachment characteristics as measured by the ECR, attachment security may fluctuate based on situational factors, which relates to the influence of extrapharmacological factors on experiences with MDMA-AT (i.e., set and setting). To address this, the Security subscale of the State Adult Attachment Measure (SAAM) will be administered. Higher scores indicate higher security in attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Harwood-Gross, PhD, Study Director — Metiv Israel Psychotrauma Center; Pinhas Danon, Prof, Principal Investigator — Herzog Medical Center
Locations (1):
- METIV Israel Psychotrauma Center, Herzog Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
Protocol is freely available along with access to data assessment plan. Data will be anonymized and available on request and uploaded to open science framework
Supporting Information: Study Protocol, SAP
Time Frame: Available currently
Access Criteria: Protocol is available to researchers on request
URL: http://www.metiv.org

REFERENCES:
- See also: Study recruitment page — https://metiv.org/sea-it-mdma/